CLINICAL TRIAL: NCT03095014
Title: Cesarean Myomectomy : Safety and Risk of Intrauterine Synechiae
Brief Title: Myomectomy During Cesarean Section
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant professor, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zuh- 5
Record Dates: First submitted 2017-03-16; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Myomectomy
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Intervention Model Description: Cesarean Myomectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cesarean Myomectomy (Experimental): Myomectomy plus Cesarean section
  Interventions: Procedure: Cesarean Myomectomy
- Cesarean section (Active Comparator): Cesarean section only
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: Cesarean Myomectomy — Myomectomy was done during Cesarean section
  Arms: Cesarean Myomectomy
Procedure: Cesarean section — Cesarean delivery
  Arms: Cesarean section

SUMMARY:
Cesarean Myomectomy, safety and effect on uterine cavity.

DETAILED DESCRIPTION:
this study aims to compare between women who underwent Cesarean Myomectomy and those who underwent Cesarean section only regarding the procedure safety and whether uterine cavity was affected later on.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* full term
* had uterine myoma

Exclusion Criteria:

* history of coagulation disorder
* antepartum hemorrhage
* previous myomectomy
* where additional operative procedures were performed

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mean change in Haemoglobin in gm/dl | 24 hours
  pre-operative Haemoglobin minus post-operative Haemoglobin level

SECONDARY OUTCOMES:
Duration of operation in hours | 2 hours
  time to complete the procedure
intrauterine adesion adhesions | 3 months
  presence of uterine cavity adhesions

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim A el sharkwy, Principal Investigator — Zagazig University

IPD SHARING:
Plan to Share IPD: No